CLINICAL TRIAL: NCT05786521
Title: The Effect of GLP1 Receptor Agonists on Physical Function, Body Composition, and Biomarkers of Aging in Older Overweight/Obese Adults With Insulin Resistance
Brief Title: Effect of GLP1 Receptor Agonists on Physical Function, Body Composition, and Markers of Aging in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tiffany Cortes, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20220256HU; 5P30AG044271-08 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Aging; Diabetes Mellitus, Type 2; PreDiabetes; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide and lifestyle intervention (Experimental): Participants will meet with a dietician throughout the study to discuss lifestyle counseling based on recommendation in the diabetes prevention program. They will also be given semaglutide for 20 weeks.
  Interventions: Drug: Semaglutide Injectable Product; Behavioral: Lifestyle Counseling
- Lifestyle intervention (Active Comparator): Participants will meet with a dietician throughout the study to discuss lifestyle counseling based on recommendation in the diabetes prevention program
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Semaglutide will be started at 0.25mg once a week for 4 weeks followed by 0.5mg once weekly for 4 weeks followed by 1.0mg once a week for 12 weeks.
  Other Names: Semaglutide and Lifestyle Counseling
  Arms: Semaglutide and lifestyle intervention
Behavioral: Lifestyle Counseling — Lifestyle Counseling will be provided throughout study intervention

SUMMARY:
Semaglutide is a medication approved by the US Food and Drug Administration (FDA) as an antihyperglycemic (a drug that reduces glucoses in those with diabetes) and for weight management. This new study will help find out what effects, semaglutide has on people who take the drug and the drug's effect on physical function, body composition, and aging.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65
* Have prediabetes or diabetes
* BMI ≥ 27.0 kg/m2
* Living independently (not in assisted living or nursing home)

Exclusion Criteria:

* Have heart disease
* Have liver disease
* Smoke

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Cortes, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortes TM, Vasquez L, Serra MC, Robbins R, Stepanenko A, Brown K, Barrus H, Campos A, Espinoza SE, Musi N. Effect of Semaglutide on Physical Function, Body Composition, and Biomarkers of Aging in Older Adults With Overweight and Insulin Resistance: Protocol for an Open-Labeled Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 13;13:e62667. doi: 10.2196/62667. PMID 39269759

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semaglutide and Lifestyle Intervention | Lifestyle Intervention
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide and Lifestyle Intervention | Lifestyle Intervention | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (4.85) | 73.4 (4.98) | 72.65 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Lean Body Mass Change
Description: Determine if there is any change in lean body mass
Time Frame: Baseline to 20 weeks
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Semaglutide and Lifestyle Intervention | Lifestyle Intervention
Number analyzed (Participants) | 10 | 10
g | -1730.6 [-3063 to -398] | -421 [-1745 to 911]

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Semaglutide and Lifestyle Intervention | Lifestyle Intervention
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide and Lifestyle Intervention (N=10) | Lifestyle Intervention (N=10)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT05786521/Prot_SAP_002.pdf
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05786521/ICF_000.pdf